CLINICAL TRIAL: NCT03186976
Title: Reversal of Atrial Substrate to Prevent Atrial Fibrillation - A Pilot Study
Brief Title: Reversal of Atrial Substrate to Prevent Atrial Fibrillation Pilot Study
Acronym: RASTA-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Cardiovascular Society (Other)
Responsible Party: Principal Investigator, Ratika Parkash, MD, FRCPC, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RP-004
Record Dates: First submitted 2017-05-31; First posted 2017-06-14 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
Keywords: Risk Factor Modification; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This will be a parallel group, open label randomized clinical trial, with blinded endpoint evaluation (PROBE design)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aggressive Risk Factor Control (Experimental): Multifaceted risk factor management relating to BP, exercise, sleep apnea, alcohol intake and diabetes management
  Interventions: Behavioral: Aggressive Risk Factor Control
- Standard of Care (Active Comparator): All patients in the control arm will receive therapies for AF as per the existing guidelines. BP, cholesterol, diabetic management will be administered as per the available guidelines.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Aggressive Risk Factor Control — 1.) Sleep apnea screening, therapy is recommended if apopnea-hypopnea (AHI) index is greater than 15, with a target index of less than 5.
  2) Counseling regarding alcohol reduction to 2 drinks/day for men, 1 drink/day for women, no binge drinking (>5 drinks at one setting).
  3) Participation in a 12 week structured, home-based exercise program and nutritional counseling. Weight reduction will be emphasized through modification of diet and exercise.
  4) An OMRON BP monitor will be supplied to each patient. A target SBP of <140/80 mm/Hg will be targeted.
  5) Smoking cessation - through local resources already established at each site 6) Management of diabetes to achieve HgA1c<6.5%
  Arms: Aggressive Risk Factor Control
Other: Standard of Care — Recommendations based on current guidelines
  Arms: Standard of Care

SUMMARY:
This is a pilot study to assess feasibility to conduct a multi-center, randomized trial to examine the effect of aggressive risk factor control and arrhythmia trigger-based intervention on the atrial substrate, which is involved in the development and maintenance of atrial fibrillation (AF).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a major health problem, with a prevalence of 0.4-1% of the population. It is associated with a six-fold risk of stroke and a two-fold increase in mortality, the main cardiac reason for death one year after presenting to the emergency department with AF is heart failure. It results in high healthcare costs, recurrent ED visits and hospitalizations. The burden of disability associated with AF has been found to increase by 20% from 1990-2010. AF was also cited as one of the seven causes of death that has been increasing worldwide. Prevention of AF has not been a focus of past treatments and it is well known that elevated body mass index, hypertension, smoking, increased alcohol intake, lack of exercise and sleep apnea are risk factors for AF. There is a lack of randomized, multicenter data proving that a strategy of aggressive risk factor modification will prevent and modify AF.

Upstream therapy for AF has been of considerable interest, and benefit has been demonstrated in primary prevention of AF. Catheter ablation has demonstrated success over current medical therapies for long-term rhythm control, but recurrence remains high, irrespective of ablation strategy. This study is a feasibility study to determine whether a complex and multi-component risk factor modification can be successfully implemented.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic (CCS-SAF ≥2) recurrent paroxysmal or persistent nonvalvular atrial fibrillation despite rate control, desiring catheter ablation AND
* one of : BMI>27, BP>140/90 or history of hypertension, alcohol use > recommended limit, current smoking, diabetes with HgA1C>7%, physical inactivity (<150 minutes/week).

(Definitions: Recurrent paroxysmal - at least 4 episodes of symptomatic AF in the prior 6 months, with or without cardioversion; Persistent AF lasting greater than 7 days but less than 3 years; AF must be documented on a Holter, rhythm strip or electrocardiogram within the last 24 months.)

Exclusion Criteria:

* Permanent AF (AF lasting > 3 years)
* Prior catheter ablation for AF
* Left ventricular ejection fraction <30%
* Left atrial size > 5.5 cm
* NYHA IV heart failure
* Participation in a cardiac rehabilitation program within the last year
* Currently performing exercise training 150 minutes/week of moderate to vigorous physical activity
* Unable to exercise
* Unable to give informed consent
* Other noncardiovascular medical condition making 1 year survival unlikely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
adherence to the risk factor intervention | 6 months
  80% compliance to each of the components: 150 minutes exercise/week, BP target as per CHEP guidelines, alcohol limits, smoking cessation, and sleep apnea therapy, hemoglobin A1C<6.5% at the end of follow up. If 80% of individuals can reach these 80% of the time, the adherence criteria will be met.

SECONDARY OUTCOMES:
Feasibility of recruitment | 6 months
  Recruitment of ≥2.8 patients/center/month over three centers, thereby completing recruitment in 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- QE II Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No